CLINICAL TRIAL: NCT03812237
Title: A Prospective, Randomized, Controlled Trial Comparing Early Weight Bearing Versus Non-Weight Bearing Following Modified Lapidus Arthrodesis
Brief Title: Early Weight Bearing Tarsometatarsal Fusion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Associates of Michigan, PC (Other)
Collaborators: Grand Rapids Medical Education Partners (Other)
Responsible Party: Principal Investigator, John G. Anderson, MD, Orthopaedic Surgeon - Foot and Ankle, Orthopaedic Associates of Michigan, PC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OAM-TMT-01
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hallux Valgus
Keywords: Lapidus Arthrodesis; Early Weight Bearing; First Tarsometatarsal Arthrodesis
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled Trial
Masking Description: Patients were blinded to treatment until their 2 week post-operative visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (EWB) Early Weight Bearing (2 Weeks Post-op) (Experimental): Subjects in the EWB group were allowed to begin bearing 50 pounds (lbs) through their hindfoot in either the boot or the short leg cast at the two-week visit. They were allowed to advance their weightbearing as tolerated by 25 lbs every four days until full weightbearing through the hindfoot was achieved.
  Interventions: Other: (EWB) Early Weight Bearing (2 Weeks Post-op)
- (SOC) Standard of Care Weight Bearing (6-8 Weeks Post-op) (No Intervention): Subjects in the SOC group were allowed to heel touch weightbear for balance only on the operative foot until the six to eight week visit. At this visit all subjects were placed into a short leg walking boot. Non-weightbearing patients were permitted to begin the progressive weightbearing protocol, without hindfoot restriction.

INTERVENTIONS:
Other: (EWB) Early Weight Bearing (2 Weeks Post-op) — Patient were permitted to progressively weightbear on their heel at 2 week post-op.
  Other Names: EWB
  Arms: (EWB) Early Weight Bearing (2 Weeks Post-op)

SUMMARY:
A Prospective, Randomized, Controlled Trial Comparing Early Weight Bearing versus Non Weight Bearing Following Modified Lapidus Arthrodesis

DETAILED DESCRIPTION:
The purpose of this prospective randomized control trial is to assess outcomes in patients who undergo modified Lapidus arthrodesis and whose postoperative management includes early weight bearing on heel (in a boot) and compare it to standard of care non weight bearing post operative management.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the Institutional Review Board approved informed consent form specific to this study prior to enrollment
* Failure of conservative treatment (i.e. non-surgical action, consisting of footwear modification in the form of shoes with wide toe boxes, padded inserts, activity modifications and pain control medications)
* Patients who underwent Lapidus procedure with or without other procedures of the first ray (i.e., muscle-tendon procedures, distal metatarsal osteotomy, Akin procedure)
* Patient older than 18 years of age
* Patient is able to give informed consent
* Patient is independent, ambulatory, and agrees to comply with all postoperative visits

Exclusion Criteria:

* Patient has a pre-existing condition which may cause impairment of healing and bone fusion
* Any significant pathology that, in the opinion of investigator, makes the patient unsuitable for study
* Patients who underwent Lapidus arthrodesis in conjunction with other procedures that did not focus on the first pedal ray with the exception of harvesting autogenous ipsilateral calcaneal bone graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
TMT Fusion Rate | 6 months
  To compare the incidence and rate of first TMT fusion using two different postoperative protocols until fusion consolidation.

SECONDARY OUTCOMES:
American Foot & Ankle Society Midfoot Scores (AOFAS) | 12 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period.] AOFAS Scale: [0 (no function/severe deformity) to 83 (full function/no limitations/deformity)]
Short Musculoskeletal Function Assessment (SMFA) | 12 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period. SMFA Scale: 101 items scored 1 to 5 [1( problems/no difficulty/not bothered) - 5 (unable to do task/symptoms constantly/extremely bothered)]
Visual Analogue Scale (VAS) | 12 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period. VAS assessment: [0 (no pain) - 10 (worse possible pain)]
Foot Function Index Revised (FFIr) | 12 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period. FFIr Scale: 67 items scored 1 to 7 [1(no problems/no difficulty/not bothered) - 6 (unable to do a task/symptoms all the time/worst pain imaginable) - 7 (Not applicable)]. Score range: 46 to 230.
Short Form Health Survey (SF-36) v.2 | 12 months
  Assessment of clinical/subjective feedback via questionnaires during the postoperative follow up period. SF-36 v.2 Scale: Self-reporting outcomes assessment [0 (no function/severe physical/mental disability) to 100 (full function, no limitations to mental/physical health)]. Score range: 46 to 230.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bednarz PA, Manoli A 2nd. Modified lapidus procedure for the treatment of hypermobile hallux valgus. Foot Ankle Int. 2000 Oct;21(10):816-21. doi: 10.1177/107110070002101004. PMID 11128011
- [Background] Clark HR, Veith RG, Hansen ST Jr. Adolescent bunions treated by the modified Lapidus procedure. Bull Hosp Jt Dis Orthop Inst. 1987 Fall;47(2):109-22. PMID 2825872
- [Background] Saxena A, Nguyen A, Nelsen E. Lapidus bunionectomy: Early evaluation of crossed lag screws versus locking plate with plantar lag screw. J Foot Ankle Surg. 2009 Mar-Apr;48(2):170-9. doi: 10.1053/j.jfas.2008.12.009. PMID 19232969
- [Background] Rutherford RL. The Lapidus procedure for primus metatarsus adductus. J Am Podiatry Assoc. 1974 Aug;64(8):581-4. doi: 10.7547/87507315-64-8-581. No abstract available. PMID 4845803
- [Background] McInnes BD, Bouche RT. Critical evaluation of the modified Lapidus procedure. J Foot Ankle Surg. 2001 Mar-Apr;40(2):71-90. doi: 10.1016/s1067-2516(01)80048-x. PMID 11324674
- [Background] Bacardi BE, Boysen TJ. Considerations for the Lapidus operation. J Foot Surg. 1986 Mar-Apr;25(2):133-8. PMID 3711593
- [Background] Christenson C, Jones RO, Basque M, Mollohan E. Comparison of oblique closing base wedge osteotomies of the first metatarsal: stripping versus nonstripping of the periosteum. J Foot Surg. 1991 Mar-Apr;30(2):107-13. PMID 1865058
- [Background] Hansen ST Jr. Hallux valgus surgery. Morton and Lapidus were right! Clin Podiatr Med Surg. 1996 Jul;13(3):347-54. PMID 8829031
- [Background] Mendicino R, Catanzariti AR, Hofbauer M, Saltrick KR. The modified lapidus arthrodesis: technical maneuvers and pearls. J Foot Ankle Surg. 2000 Jul-Aug;39(4):258-64. doi: 10.1016/s1067-2516(00)80010-1. No abstract available. PMID 10949807
- [Result] LAPIDUS PW. The author's bunion operation from 1931 to 1959. Clin Orthop. 1960;16:119-35. No abstract available. PMID 14414101
- [Result] Sangeorzan BJ, Hansen ST Jr. Modified Lapidus procedure for hallux valgus. Foot Ankle. 1989 Jun;9(6):262-6. doi: 10.1177/107110078900900602. PMID 2744666
- [Result] Myerson M, Allon S, McGarvey W. Metatarsocuneiform arthrodesis for management of hallux valgus and metatarsus primus varus. Foot Ankle. 1992 Mar-Apr;13(3):107-15. doi: 10.1177/107110079201300301. PMID 1601337
- [Result] Hernandez A, Hernandez PA, Hernandez WA. Lapidus: when and why? Clin Podiatr Med Surg. 1989 Jan;6(1):197-208. PMID 2653609
- [Result] Catanzariti AR, Mendicino RW, Lee MS, Gallina MR. The modified Lapidus arthrodesis: a retrospective analysis. J Foot Ankle Surg. 1999 Sep-Oct;38(5):322-32. doi: 10.1016/s1067-2516(99)80003-9. PMID 10553545
- [Result] Myerson MS, Badekas A. Hypermobility of the first ray. Foot Ankle Clin. 2000 Sep;5(3):469-84. PMID 11232392
- [Result] Ray RG. First metatarsocuneiform arthrodesis: technical considerations and technique modification. J Foot Ankle Surg. 2002 Jul-Aug;41(4):260-72. doi: 10.1016/s1067-2516(02)80025-4. PMID 12194518
- [Result] Kopp FJ, Patel MM, Levine DS, Deland JT. The modified Lapidus procedure for hallux valgus: a clinical and radiographic analysis. Foot Ankle Int. 2005 Nov;26(11):913-7. doi: 10.1177/107110070502601103. PMID 16309603
- [Result] Coetzee JC, Resig SG, Kuskowski M, Saleh KJ. The Lapidus procedure as salvage after failed surgical treatment of hallux valgus. Surgical technique. J Bone Joint Surg Am. 2004 Mar;86-A Suppl 1:30-6. doi: 10.2106/00004623-200403001-00005. PMID 14996919
- [Result] Saffo G, Wooster MF, Stevens M, Desnoyers R, Catanzariti AR. First metatarsocuneiform joint arthrodesis: a five-year retrospective analysis. J Foot Surg. 1989 Sep-Oct;28(5):459-65. PMID 2584630
- [Result] Gutteck N, Wohlrab D, Zeh A, Radetzki F, Delank KS, Lebek S. Immediate fullweightbearing after tarsometatarsal arthrodesis for hallux valgus correction--Does it increase the complication rate? Foot Ankle Surg. 2015 Sep;21(3):198-201. doi: 10.1016/j.fas.2014.11.010. Epub 2014 Dec 29. PMID 26235860
- [Result] Goldstein CL, Schemitsch E, Bhandari M, Mathew G, Petrisor BA. Comparison of different outcome instruments following foot and ankle trauma. Foot Ankle Int. 2010 Dec;31(12):1075-80. doi: 10.3113/FAI.2010.1075. PMID 21189208
- [Result] Prissel MA, Hyer CF, Grambart ST, Bussewitz BW, Brigido SA, DiDomenico LA, Lee MS, Reeves CL, Shane AM, Tucker DJ, Weinraub GM. A Multicenter, Retrospective Study of Early Weightbearing for Modified Lapidus Arthrodesis. J Foot Ankle Surg. 2016 Mar-Apr;55(2):226-9. doi: 10.1053/j.jfas.2015.09.003. Epub 2016 Jan 5. PMID 26763868
- [Result] King CM, Richey J, Patel S, Collman DR. Modified lapidus arthrodesis with crossed screw fixation: early weightbearing in 136 patients. J Foot Ankle Surg. 2015 Jan-Feb;54(1):69-75. doi: 10.1053/j.jfas.2014.09.034. Epub 2014 Oct 31. PMID 25451208